CLINICAL TRIAL: NCT01371708
Title: A 6-month, Open-label, Multi-center, Flexible Dose Extension Study To The B2061032 Study To Evaluate The Safety, Tolerability And Efficacy Of Desvenlafaxine Succinate Sustained Release (Dvs Sr) Tablets In The Treatment Of Children And Adolescent Outpatients With Major Depressive Disorder
Brief Title: A 6-Month Extension Study To The B2061032 Study To Evaluate The Safety, Tolerability, And Efficacy Of DVS SR In The Treatment Of Child And Adolescent Outpatients With MDD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2061030; 3151A6-3344 (Other: Alias Study Number); 2008-001876-67 (EudraCT Number)
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Desvenlafaxine Succinate Sustained-Release (Experimental)
  Interventions: Drug: DVS SR

INTERVENTIONS:
Drug: DVS SR — Subjects will receive a flexible-dose of 20, 25, 35, or 50 mg/day as prescribed by the investigator

SUMMARY:
This is a 6-month, open-label, flexible-dose study evaluating Desvenlafaxine Succinate Sustained-Release (DVS SR) in the Treatment of Child and Adolescent Outpatients with Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Completed study B2061032 and who in the investigator's opinion, would benefit from long term treatment with DVS SR
* Willingness and ability to comply with scheduled visits, treatment plan, and procedures

Exclusion Criteria:

* Requires precaution against suicide
* Not in generally healthy medical condition
* Poor compliance with study drug or study procedures during participation in study B2061032

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 283 (Actual)
Dates: Start 2012-02-02 (Actual); Primary Completion 2016-04-22 (Actual); Study Completion 2016-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- United States (35):
  - The University Of Alabama At Birmingham, Office Of Psychiatric Research, Birmingham, Alabama
  - Center for Advanced Improvement, Tucson, Arizona
  - Sun Valley Research Center, Imperial, California
  - MCB Clinical Research Centers, Colorado Springs, Colorado
  - Institute of Living/Hartford Hospital, Hartford, Connecticut
  - SJS Clinical Research, Inc., Destin, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Jacksonville, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Millenia Psychiatry & Research, Inc., Orlando, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - Baber Research Group, Naperville, Illinois
  - Clinco, Terre Haute, Indiana
  - Pharmasite Research, Inc, Baltimore, Maryland
  - Millennium Psychiatric Associates, LLC, Creve Coeur, Missouri
  - Premier Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - Erie County Medical Center/State University of New York (SUNY) at Buffalo Affiliate, Buffalo, New York
  - The Zucker Hillside Hospital, North Shore-Long Island Jewish Health System, Glen Oaks, New York
  - Bioscience Research, LLC., Mount Kisco, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Stony Brook University Medical Center, child and Adolescent Psychiatry, Stony Brook, New York
  - Neuro-Behavioral Clinical Research, Inc., Canton, Ohio
  - Discovery and Wellness Center for Children/University Hospitals Case Medical Center, Cleveland, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Research Strategies of Memphis, LLC., Memphis, Tennessee
  - FutureSearch Trials, Austin, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Clinical Trials of Texas, INC, San Antonio, Texas
  - Allance Research Group, Richmond, Virginia
  - Alliance Research Group, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Treatment Center for Children, Richmond, Virginia
  - Eastside Therapeutic Resource, Kirkland, Washington
- Biomedica Research Group, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Derived] Atkinson S, Thurman L, Ramaker S, Buckley G, Jones SR, England R, Wajsbrot D. Safety, Tolerability, and Efficacy of Desvenlafaxine in Children and Adolescents with Major Depressive Disorder: Results from Two Open-Label Extension Trials. CNS Spectr. 2019 Oct;24(5):496-506. doi: 10.1017/S1092852918001128. PMID 30419989
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2061030&StudyName=A%206-Month%20Extension%20Study%20To%20The%20B2061032%20Study%20To%20Evaluate%20The%20Safety%2C%20Tolerability%2C%20And%20Efficacy%20Of%20DVS%20SR%20In%20The%20Treatment%20Of

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 304 participants completed study B2061032, 283 of whom were enrolled in the current extension study, B2061030, and 281 received treatment.
Groups:
- Placebo/DVS-SR: Participants received placebo tablets in previous study B2061032 and desvenlafaxine succinate sustained-release (DVS-SR) in flexible dosing ranging from 20 to 50 mg in extension study B2061030.
- DVS-SR, Low Dose/DVS-SR: Participants received DVS-SR in weight-based dosing (20, 25, or 35 mg) in previous study B2061032, and DVS-SR in flexible dosing ranging from 20 to 50 mg in extension study B2061030.
- DVS-SR, High Dose/DVS-SR: Participants received DVS-SR in weight-based dosing (25, 35, or 50 mg) in previous study B2061032, and DVS-SR in flexible dosing ranging from 20 to 50 mg in extension study B2061030.
Period: Overall Study
Arm/Group | Placebo/DVS-SR | DVS-SR, Low Dose/DVS-SR | DVS-SR, High Dose/DVS-SR
Started | 92 | 93 | 98
Received Treatment | 91 | 93 | 97
Completed | 66 | 63 | 59
Not Completed | 26 | 30 | 39
Not completed — Insufficient clinical response | 3 | 2 | 0
Not completed — Lost to Follow-up | 5 | 9 | 7
Not completed — Protocol Violation | 2 | 1 | 2
Not completed — No longer willing to participate | 7 | 7 | 13
Not completed — Medication error/not related to AE | 0 | 1 | 0
Not completed — Other | 3 | 2 | 4
Not completed — Adverse Event | 5 | 8 | 12
Not completed — Started but did not receive treatment | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/DVS-SR | DVS-SR, Low Dose/DVS-SR | DVS-SR, High Dose/DVS-SR | Total
Number analyzed (Participants) | 91 | 93 | 97 | 281
Age, Customized [Number; unit: Participants]
  7 to 11 years | 28 | 26 | 33 | 87
  12 to 17 years | 63 | 67 | 64 | 194
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 52 | 60 | 155
  Male | 48 | 41 | 37 | 126
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 1 | 0 | 2
  Black or African American | 20 | 23 | 28 | 71
  White | 62 | 65 | 60 | 187
  Other | 8 | 4 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as an event that was absent before treatment and emerged or worsened during the treatment period.
Time Frame: From Week 8 (B2061032)/Day 1 (B2061030) to Week 26 of B2061030
Population: All participants who received at least 1 dose of study drug in study B2061030
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo/DVS-SR | DVS-SR, Low Dose/DVS-SR | DVS-SR, High Dose/DVS-SR
Number analyzed (Participants) | 91 | 93 | 97
Percentage of participants | 78.0 | 73.1 | 71.1

2. Primary Outcome: Percentage of Participants With a Treatment-emergent Adverse Event (TEAE) (Combination Group)
Description: A TEAE was defined as an event that was absent before treatment and emerged or worsened during the treatment period.
Time Frame: From Week 8 (B2061032)/Day 1 (B2061030) to Week 26 of B2061030
Population: All participants who received at least 1 dose of study drug in study B2061030
Measure: Number; unit: Percentage of participants
Groups:
- Combination Group: Combination of 3 groups of participants from previous study B2061032 received desvenlafaxine succinate sustained release in flexible dosing ranging from 20 to 50 mg in the current extension study, B2061030.
Arm/Group | Combination Group
Number analyzed (Participants) | 281
Percentage of participants | 74.0

3. Secondary Outcome: Change From Baseline to Week 26 in Total Score on the Children's Depression Rating Scale, Revised (CDRS-R), Based on Observed Cases
Description: The CDRS-R consists of 17 items. The total score is the sum of responses to the 17 items and ranges from 17 to 113. Lower total scores indicate lower intensity of symptoms. Remission on the CDRS-R was defined as a CDRS-R score <=28. It was recommended that the CDRS-R be performed prior to the Clinical Global Impression assessments. Mean change from baseline=score at Week 26 minus score at baseline of study B2061032.
Time Frame: From Week 8 (B2061032)/Day 1 (B2061030) to Week 26 of B2061030
Population: All participants who had a CDRS-R evaluation at Baseline of study B2061030 (Week 8 of study B2061032), took at least 1 dose of study drug, and had at least 1 CDRS-R evaluation after the first dose of study drug in B2061030.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo/DVS-SR | DVS-SR, Low Dose/DVS-SR | DVS-SR, High Dose/DVS-SR
Number analyzed (Participants) | 63 | 57 | 56
Units on a scale | -6.79 (12.05) | -10.72 (10.80) | -8.57 (13.01)

4. Secondary Outcome: Change From Baseline to Week 26 in Total Score on the Children's Depression Rating Scale, Revised (CDRS-R), Based on Observed Cases (Combination Group)
Description: as for outcome 3
Time Frame: From Week 8 (B2061032)/Day 1 (B2061030) to Week 26 of B2061030
Population: All participants who had a CDRS-R evaluation at Baseline of study B2061030 (Week 8 of study B2061032), took at least 1 dose of study drug, had at least 1 CDRS-R evaluation after the first dose of study drug in B2061030, and were available for evaluation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Combination Group
Number analyzed (Participants) | 176
Units on a scale | -8.63 (12.03)

5. Secondary Outcome: Change in Score From Baseline to Week 26 on the Clinical Global Impression-Severity (CGI-S) Scale, Based on Observed Cases
Description: The Clinical Global Impression (CGI) Scale is a tool that summarizes all available patient data, including history, symptoms, behavior, and the impact of the symptoms on ability to function. The scale consists of 2 measures: the CGI-S, which rates the severity of illness from 1 to 7, and the CGI-Improvement Scale, which assesses improvement in illness since baseline. The CGI-S is a 7-point scale a clinician uses to rate a patient's severity of illness. Scores range from 1 to 7, with 1 indicating "normal, not at all ill" and 7, "among the most extremely ill patients." Higher score on the CGI-S indicates greater severity of illness. Mean change from baseline=score at Week 26 minus score at baseline of study B2061032.
Time Frame: From Week 8 (B2061032)/Day 1 (B2061030) to Week 26 of B2061030
Population: All participants who had a Children's Depression Rating Scale-Revised (CDRS-R) evaluation at Baseline of study B2061030 (Week 8 of study B2061032), took at least 1 dose of study drug, and had at least 1 CDRS-R evaluation after the first dose of study drug in B2061030.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo/DVS-SR | DVS-SR, Low Dose/DVS-SR | DVS-SR, High Dose/DVS-SR
Number analyzed (Participants) | 63 | 57 | 56
Units on a scale | -1.02 (1.18) | -1.44 (1.12) | -0.70 (1.37)

6. Secondary Outcome: Change in Score From Baseline to Week 26 on the Clinical Global Impression-Severity (CGI-S) Scale, Based on Observed Cases (Combination Group)
Description: as for outcome 5
Time Frame: From Week 8 (B2061032)/Day 1 (B2061030) to Week 26 of B2061030
Population: All participants who had a Children's Depression Rating Scale-Revised (CDRS-R) evaluation at Baseline of study B2061030 (Week 8 of study B2061032), took at least 1 dose of study drug, had at least 1 CDRS-R evaluation after the first dose of study drug in B2061030, and were available for evaluation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Combination Group
Number analyzed (Participants) | 176
Units on a scale | -1.05 (1.26)

7. Secondary Outcome: Percentage of Participants With a Response of Very Much Improved or Much Improved on the Clinical Global Impression-Improvement (CGI-I) Scale at Week 26, Based on Observed Cases
Description: The Clinical Global Impression (CGI) Scale is a tool that summarizes all available patient data, including history, symptoms, behavior, and the impact of the symptoms on ability to function. The scale consists of 2 measures: the CGI-Severity scale, which rates the severity of illness from 1 to 7, and the CGI-I scale, which assesses improvement in illness since baseline. The CGI-I is a 7-point scale a clinician uses to assess improvement in a patient's illness relative to baseline. Scores range from 1 to 7, with 1 representing "very much improved" and 7 representing "very much worse"; a value of 0 meant not assessed. Lower score indicates greater improvement. Response on the CGI-I defined as the CGI-I scores of 1 or 2. Mean change from baseline=score at Week 26 minus score at baseline of study B2061032.
Time Frame: From Week 8 (B2061032)/Day 1 (B2061030) to Week 26 of B2061030
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo/DVS-SR | DVS-SR, Low Dose/DVS-SR | DVS-SR, High Dose/DVS-SR
Number analyzed (Participants) | 63 | 57 | 56
Percentage of participants | 87.3 | 94.7 | 89.3

8. Secondary Outcome: Percentage of Participants With a Response of Very Much Improved or Much Improved on the Clinical Global Impression-Improvement (CGI-I) Scale at Week 26, Based on Observed Cases (Combination Group)
Description: as for outcome 7
Time Frame: From Week 8 (B2061032)/Day 1 (B2061030) to Week 26 of B2061030
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Combination Group
Number analyzed (Participants) | 176
Percentage of participants | 90.3

9. Secondary Outcome: Percentage of Participants by Score on the Clinical Global Impression-Improvement (CGI-I) Scale, Based on Observed Cases
Description: The Clinical Global Impression (CGI) Scale is a tool that summarizes all available patient data, including history, symptoms, behavior, and the impact of the symptoms on ability to function. The scale consists of 2 measures: the CGI-Severity scale, which rates the severity of illness from 1 to 7, and the CGI-I scale, which assesses improvement in illness since baseline. The CGI-I is a 7-point scale used a clinician uses to assess improvement in a patient's illness relative to baseline. Scores range from 1 to 7, with 1 representing "very much improved" and 7 representing "very much worse"; a value of 0 meant not assessed. Lower score indicates greater improvement. Response on the CGI-I defined as the CGI-I scores of 1 or 2. Mean change from baseline=score at Week 26 minus score at baseline of study B2061032.
Time Frame: From Week 8 (B2061032)/Day 1 (B2061030) to Week 26 of B2061030
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo/DVS-SR | DVS-SR, Low Dose/DVS-SR | DVS-SR, High Dose/DVS-SR
Number analyzed (Participants) | 63 | 57 | 56
Percentage of participants
  Week 26: Very much improved | 54.0 | 73.7 | 53.6
  Week 26: Much improved | 33.3 | 21.1 | 35.7
  Week 26: Minimally improved | 9.5 | 5.3 | 10.7
  Week 26: No change | 1.6 | 0.0 | 0.0
  Week 26: Minimally worse | 1.6 | 0.0 | 0.0
  Week 26: Much worse | 0.0 | 0.0 | 0.0
  Week 26: Very much worse | 0.0 | 0.0 | 0.0

10. Secondary Outcome: Percentage of Participants by Score on the Clinical Global Impression-Improvement (CGI-I) Scale, Based on Observed Cases (Combination Group)
Description: as for outcome 9
Time Frame: From Week 8 (B2061032)/Day 1 (B2061030) to Week 26 of B2061030
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Combination Group
Number analyzed (Participants) | 176
Percentage of participants
  Week 26: Very much improved | 60.2
  Week 26: Much improved | 30.1
  Week 26: Minimally improved | 8.5
  Week 26: No change | 0.6
  Week 26: Minimally worse | 0.6
  Week 26: Much worse | 0.0
  Week 26: Very much worse | 0.0

11. Secondary Outcome: Percentage of Participants With Remission at Week 26, Based on Score on the Children's Depression Rating Scale, Revised (CDRS-R), <=28 and on Observed Cases
Description: Remission on the CDRS-R was defined as a CDRS-R score <=28. The CDRS-R consists of 17 items. The total score is the sum of responses to the 17 items and ranges from 17 to 113. Lower total s cores indicate lower intensity of symptoms.
Time Frame: From Week 8 (B2061032)/Day 1 (B2061030) to Week 26 of B2061030
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo/DVS-SR | DVS-SR, Low Dose/DVS-SR | DVS-SR, High Dose/DVS-SR
Number analyzed (Participants) | 63 | 57 | 56
Percentage of participants | 73.0 | 89.5 | 75.0

12. Secondary Outcome: Percentage of Participants With Remission at Week 26, Based on a Score on the Children's Depression Rating Scale, Revised (CDRS-R), <=28 and on Observed Cases (Combination Group)
Description: as for outcome 11
Time Frame: From Week 8 (B2061032)/Day 1 (B2061030) to Week 26 of B2061030
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Combination Group
Number analyzed (Participants) | 176
Percentage of participants | 79.0

ADVERSE EVENTS:
Time Frame: From informed consent through Week 30 (adverse events) and Week 32 visit (serious adverse events). For participants who discontinued prior to Week 28 visit: Adverse events collected for 14 days, and serious adverse events for 28 days,
Groups:
- DVS-SR, Low Dose/DVS-SR: Participants received DVS-SR in weight-based dosing(20, 25, or 35 mg) in previous study B2061032, and DVS-SR in flexible dosing ranging from 20 to 50 mg in extension study B2061030.
- Combination Group: Combination of 3 groups of participants from previous study B2061032 received DVS-SR in flexible dosing ranging from 20 to 50 mg in extension study B2061030.
Arm/Group | Placebo/DVS-SR | DVS-SR, Low Dose/DVS-SR | DVS-SR, High Dose/DVS-SR | Combination Group
Serious Adverse Events (participants affected / at risk) | 4/91 | 6/93 | 3/97 | 13/281
Other Adverse Events (participants affected / at risk) | 60/91 | 57/93 | 58/97 | 175/281
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/DVS-SR (N=91) | DVS-SR, Low Dose/DVS-SR (N=93) | DVS-SR, High Dose/DVS-SR (N=97) | Combination Group (N=281)
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 1 | 0 | 2
Hallucination, auditory (Psychiatric disorders) | 0 | 1 | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 1
Pyromania (Psychiatric disorders) | 0 | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 1 | 2 | 5
Suicide attempt (Psychiatric disorders) | 0 | 2 | 1 | 3
Suicide threat (Psychiatric disorders) | 1 | 0 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/DVS-SR (N=91) | DVS-SR, Low Dose/DVS-SR (N=93) | DVS-SR, High Dose/DVS-SR (N=97) | Combination Group (N=281)
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1 | 8 | 13
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 5 | 8
Nausea (Gastrointestinal disorders) | 4 | 11 | 6 | 21
Vomiting (Gastrointestinal disorders) | 6 | 2 | 4 | 12
Fatigue (General disorders) | 3 | 0 | 3 | 6
Gastroenteritis (Infections and infestations) | 3 | 2 | 1 | 6
Gastroenteritis viral (Infections and infestations) | 7 | 3 | 6 | 16
Nasopharyngitis (Infections and infestations) | 9 | 4 | 8 | 21
Otitis media (Infections and infestations) | 3 | 1 | 1 | 5
Pharyngitis streptococcal (Infections and infestations) | 1 | 1 | 3 | 5
Sinusitis (Infections and infestations) | 1 | 2 | 5 | 8
Upper respiratory tract infection (Infections and infestations) | 4 | 10 | 2 | 16
Accidental overdose (Injury, poisoning and procedural complications) | 8 | 4 | 8 | 20
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 3
Weight increased (Investigations) | 5 | 4 | 5 | 14
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 1 | 7
Increased appetite (Metabolism and nutrition disorders) | 0 | 3 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 7
Dizziness (Nervous system disorders) | 4 | 6 | 5 | 15
Headache (Nervous system disorders) | 12 | 16 | 17 | 45
Psychomotor hyperactivity (Nervous system disorders) | 3 | 1 | 0 | 4
Somnolence (Nervous system disorders) | 10 | 3 | 1 | 14
Agitation (Psychiatric disorders) | 0 | 2 | 3 | 5
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 3 | 1 | 2 | 6
Depression (Psychiatric disorders) | 1 | 3 | 4 | 8
Initial insomnia (Psychiatric disorders) | 5 | 0 | 1 | 6
Insomnia (Psychiatric disorders) | 7 | 6 | 4 | 17
Irritability (Psychiatric disorders) | 3 | 4 | 7 | 14
Self injurious behaviour (Psychiatric disorders) | 0 | 3 | 1 | 4
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 3 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.